CLINICAL TRIAL: NCT04549883
Title: Low Back Motor Control in Rhythmic Gymnasts During Hip Extension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Maria Fortun Agud, Principal Investigator, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LBcontrolGymnasts
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Low Back Pain
Keywords: gymnastics; low back pain; Physical Therapy Specialty
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: single-group, pretest-posttest clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Performing after session (Experimental): LB control during hip extension after intervention
  Interventions: Other: Theoretical practical educational session

INTERVENTIONS:
Other: Theoretical practical educational session — 1 Theoretical practical educational session of 15 Min about the importance of low back control during hip extension. Includes anatomical issues and one practical exercise in quadruped position

SUMMARY:
CONTEXT: Low back pain (LBP) is a common complaint in gymnasts. A deficit in the control of lumbopelvic movement has been related to low back pain. OBJECTIVE: This study aims to examine the effectiveness of an education session about low back motor control during hip extension in the lumbopelvic sagittal movement control of elite gymnasts.

DESIGN: single-group, pretest-posttest clinical trial. PARTICIPANTS: 70 Elite Rhythmic Gymnasts INTERVENTION: One standardized theoretical practical session of 15 Min that includes anatomical issues and one practical exercise in quadruped position for controlling the movement of lumbar spine during hip extension and flexion.

ELIGIBILITY:
Inclusion Criteria:

* pre-established level of practice: minimum 13 hours
* taking part in the Italian federal championship
* sign an informed consent form

Exclusion Criteria:

* not fulfill Inclusion Criteria
* had surgery in the low back pain or the hip joint

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-11-10 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Pre- spinal movement control in 10º of hip extension | Min 0 - Min 15
  Preintervention movement control of the spine in 10º of hip extension
Post- spinal movement control in 10º of hip extension | Min 30 - Min 45
  Postintervention movement control of the spine in 10º of hip extension

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fortun Agud, PhD, Principal Investigator — Unidad de Investigación en Fisioterapia Universidad de Zaragoza
Locations (1):
- Unidad de Investigación en Fisioterapia. Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Share per email to specialized manual physical therapists
Supporting Information: Study Protocol
Time Frame: 15.09.20 - 30.09.20
Access Criteria: email

REFERENCES:
- [Result] Sweeney EA, Daoud AK, Potter MN, Ritchie L, Howell DR. Association Between Flexibility and Low Back Pain in Female Adolescent Gymnasts. Clin J Sport Med. 2019 Sep;29(5):379-383. doi: 10.1097/JSM.0000000000000660. PMID 31460951
- [Result] Crasto CFB, Montes AM, Carvalho P, Carral JMC. Pressure biofeedback unit to assess and train lumbopelvic stability in supine individuals with chronic low back pain. J Phys Ther Sci. 2019 Oct;31(10):755-759. doi: 10.1589/jpts.31.755. Epub 2019 Oct 19. PMID 31645801
- [Result] Ramos LAV, Callegari B, Franca FJR, Magalhaes MO, Burke TN, Carvalho E Silva APMC, Almeida GPL, Comachio J, Marques AP. Comparison Between Transcutaneous Electrical Nerve Stimulation and Stabilization Exercises in Fatigue and Transversus Abdominis Activation in Patients With Lumbar Disk Herniation: A Randomized Study. J Manipulative Physiol Ther. 2018 May;41(4):323-331. doi: 10.1016/j.jmpt.2017.10.010. PMID 29751850
- [Result] Azevedo DC, Lauria AC, Pereira AR, Andrade GT, Ferreira ML, Ferreira PH, Van Dillen L. Intraexaminer and interexaminer reliability of pressure biofeedback unit for assessing lumbopelvic stability during 6 lower limb movement tests. J Manipulative Physiol Ther. 2013 Jan;36(1):33-43. doi: 10.1016/j.jmpt.2012.12.008. PMID 23380212
- [Result] Fawcett L, Heneghan NR, James S, Rushton A. Perceptions of low back pain in elite gymnastics: A multi-disciplinary qualitative focus group study. Phys Ther Sport. 2020 Jul;44:33-40. doi: 10.1016/j.ptsp.2020.04.003. Epub 2020 Apr 18. PMID 32375075